CLINICAL TRIAL: NCT01829269
Title: French Attitude Registry in Case of ICD Lead Replacement
Acronym: FRAGILE
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 12 759
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Defibrillator; Explantation of Probe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a defibrillator: The study population is that of patients with a defibrillator to have a change of probe.

SUMMARY:
The average survival rate of a defibrillation lead is 91 to 99% at 2 years, 85-95% at 5 years and 60-72% at 8 years. We must also manage alerts for defibrillation probes with a higher complication rate than average. We will therefore be increasingly confronted with faulty sensors or at risk to be replaced.

There are no standardized approach for replacing defibrillation lead. A record made in the United States showed significant differences according to the teams strategy in case of failure of defibrillation lead in particular with regard to the decision to explant or abandon the probe.

The risk of extracting a defibrillation lead are well known with a major complication rate of 1.6 to 1.95%.

Regarding the risk of complications related to the abandonment of a probe we have less data. For some there is no risk to abandon a defibrillation lead. But others reported a complication rate of 5.5% related to pacing discontinued.

Main objective: Collect the attitude of different centers and different operators when replacing a failed defibrillation lead or "at risk." Explantation or abandonment of the sensor replaced.

ELIGIBILITY:
Inclusion Criteria:

* Patient to receive a replacement defibrillation lead not motivated by an infection and having been informed.
* Patient who agreed to participate in the study
* Patients aged 18 years and over

No Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Centers are hospitals recruiters French public or private, authorized to ask defibrillators and who agreed to participate in the study. A cardiologist referral will be designated for each hospital.
  Patients with a defibrillator will be recruited during their hospitalization for change probe. Patients will receive full information about the purpose and conduct of the study.
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Explanted probes | 2 years
  Percentage of explanted probes among implanted ones

SECONDARY OUTCOMES:
Complications of explantation | 2 years
  Percentage of events during and after explantation of probe

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Ambroise Paré, Neuilly-sur-Seine, France

REFERENCES:
- [Background] Goette A, Cantu F, van Erven L, Geelen P, Halimi F, Merino JL, Morgan JM; Scientific Initiative Committee of the European Heart Rhythm Association. Performance and survival of transvenous defibrillation leads: need for a European data registry. Europace. 2009 Jan;11(1):31-4. doi: 10.1093/europace/eun301. Epub 2008 Nov 11. PMID 19004838
- [Background] Wilkoff BL, Love CJ, Byrd CL, Bongiorni MG, Carrillo RG, Crossley GH 3rd, Epstein LM, Friedman RA, Kennergren CE, Mitkowski P, Schaerf RH, Wazni OM; Heart Rhythm Society; American Heart Association. Transvenous lead extraction: Heart Rhythm Society expert consensus on facilities, training, indications, and patient management: this document was endorsed by the American Heart Association (AHA). Heart Rhythm. 2009 Jul;6(7):1085-104. doi: 10.1016/j.hrthm.2009.05.020. Epub 2009 May 22. No abstract available. PMID 19560098
- [Background] Xu W, Moore HJ, Karasik PE, Franz MR, Singh SN, Fletcher RD. Management strategies when implanted cardioverter defibrillator leads fail: survey findings. Pacing Clin Electrophysiol. 2009 Sep;32(9):1130-41. doi: 10.1111/j.1540-8159.2009.02454.x. PMID 19719488
- [Background] Rickard J, Wilkoff BL. Extraction of implantable cardiac electronic devices. Curr Cardiol Rep. 2011 Oct;13(5):407-14. doi: 10.1007/s11886-011-0198-x. PMID 21748302
- [Background] Wilkoff BL, Byrd CL, Love CJ, Hayes DL, Sellers TD, Schaerf R, Parsonnet V, Epstein LM, Sorrentino RA, Reiser C. Pacemaker lead extraction with the laser sheath: results of the pacing lead extraction with the excimer sheath (PLEXES) trial. J Am Coll Cardiol. 1999 May;33(6):1671-6. doi: 10.1016/s0735-1097(99)00074-1. PMID 10334441
- [Background] Glikson M, Suleiman M, Luria DM, Martin ML, Hodge DO, Shen WK, Bradley DJ, Munger TM, Rea RF, Hayes DL, Hammill SC, Friedman PA. Do abandoned leads pose risk to implantable cardioverter-defibrillator patients? Heart Rhythm. 2009 Jan;6(1):65-8. doi: 10.1016/j.hrthm.2008.10.012. Epub 2008 Oct 11. PMID 19121802
- [Background] Suga C, Hayes DL, Hyberger LK, Lloyd MA. Is there an adverse outcome from abandoned pacing leads? J Interv Card Electrophysiol. 2000 Oct;4(3):493-9. doi: 10.1023/a:1009860514724. PMID 11046188
- See also: Related Info — http://www.sfcardio.fr